CLINICAL TRIAL: NCT03689205
Title: Assessment of the Effect of Obesity on Venous Puncture Pain
Brief Title: The Effect of Obesity on Venous Puncture Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assist. Prof, Tokat Gaziosmanpasa University
Other Study IDs: 18-KAEK-101
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Pain; Cannulation; Body Mass Index
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients that BMI> 30kg / m2 (Group A): Venous puncture pain on patients that Body mass index > 30kg / m2
- Patients that BMI< 30kg / m2 (Group B): Venous puncture pain on patients that Body mass index < 30kg / m2

SUMMARY:
Before surgery, patients will fill the Beck anxiety, distress tolerance test and Pain katastrophizing test. Patients will be divided into two groups according to BMI> 30kg / m2 (Group A) and BMI <30kg / m2 (Group B). Compared to body weight, venous vascular pain of the groups will be compared.

DETAILED DESCRIPTION:
Seventy patients will be randomized to two groups(BMI> 30kg / m2 (Group A) and BMI <30kg / m2 (Group B) during peripheral venous cannulation (PVC). The patients' visual analog scores will be measured during peripheral venous cannulation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status 1 and 2, between the ages of 18 and 65, were scheduled for elective surgery

Exclusion Criteria:

* Patients with a history of anxiety disorders or hearing problem and preoperative pain, emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2018-11-20 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | one month
  pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)